CLINICAL TRIAL: NCT07195448
Title: The GRACE Study - Global Research on Appearance in Cancer
Brief Title: Global Research on Appearance in Cancer (GRACE)
Acronym: GRACE
Status: Recruiting | Type: Observational
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Charlotte Goodrose-Flores, RDN, PhD, Karolinska Institutet
Other Study IDs: GRACE
Record Dates: First submitted 2025-09-04; First posted 2025-09-26 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Gaining insight into how weight loss is perceived by persons with advanced cancer, and identifying potential differences related to gender and country of residence, is essential for developing comprehensive, equitable, gender-sensitive recommendations for medical nutrition therapy, with the aim of improving disease outcome.

DETAILED DESCRIPTION:
This is a multi-country cross-sectional study. Fifty men and 50 women, 18 years and above, diagnosed with advanced cancer, with a life expectancy of > 3 months, from eight countries (Australia, Chile, Germany, New Zealand, Sweden, Switzerland, USA, Vietnam) will be invited to participate. Study participants will be recruited at cancer clinics, where they will receive a QR code providing access a digital questionnaire one time. No personal information, such as name, address, or social security number, is collected. Therefore, the digital questionnaire is anonymous. Data will be collected on various variables, including weight (in kilograms or pounds) and weight history (weight before diagnosis), height (in centimeters or inches), previous weight loss attempts, education (completed high school/completed college), marital status, body image (Body Image Scale, nutrition impact symptoms (Edmonton Symptom Assessment Scale) and dietary habits (questions about choice of foods in the past week).

Regarding missing data, Body Image Scale (BIS), missing items will be handled strictly according to the scoring protocol. No imputation will be applied to other variables, which will be analyzed using complete cases.

The proposed sample size is considered appropriate and sufficient to generate valuable insights for the research community in the field of palliative care. While the sample size is not derived from a formal power calculation, the inclusion of 50 men and 50 women from each study site is anticipated to provide robust and meaningful data to address the study objectives effectively.The data will be processed at Karolinska Institutet, Stockholm, Sweden.

The statistical analysis to address the objectives is ANCOVA, which will be applied to assess group differences while controlling for covariates.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of cancer
* Must be able to understand the consent form

Exclusion Criteria:

- Expected survival time < 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Persons diagnosed with cancer.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2025-02-10 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Body image | 2025-2027
  The primary outcome measure of the GRACE study is to measure body image, by using Body Image Scale (BIS). The scoring model contains of four possible responses computing a maximum summary score of 21. The possible responses range from "not at all" (0 points) to "very much" (3 points). A higher score indicate a more distressed body image.

SECONDARY OUTCOMES:
Body Image, weight loss, percent weight loss and appetite | 2025-2027
  Weight loss measured in kilograms and percent lost compared to weight prior to cancer diagnosis.
  Appetite measured by using Edmonton Symptom Assessment Scale (ESAS). Appetite is rated between 0 (best possible appetite) to 10 (no appetite).

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska Institutet, Stockholm, Sweden